CLINICAL TRIAL: NCT02052271
Title: Thérapeutique expérimentale du Tremblement Essentiel Par la Stimulation Transcranienne Par Courant Direct (tDCS) du Cortex Cerebelleux
Brief Title: Experimental Therapeutics in Essential Tremor Using Cerebellar Transcranial Direct Current Stimulation
Acronym: ELECTRE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: C13-24; 2013-A01404-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Essential Tremor
Keywords: essential tremor; cerebellum; transcranial direct current stimulation; electrophysiology
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Essential tremor (Experimental): cerebellar stimulation
  Interventions: Device: Cathodal cerebellar transcranial direct current stimulation
- Placebo arm (Placebo Comparator): placebo stimulation
  Interventions: Device: Cathodal cerebellar transcranial direct current stimulation

INTERVENTIONS:
Device: Cathodal cerebellar transcranial direct current stimulation — Active stimulation: duration: 20 mn, intensity: 2 mA; localisation : cerebellum; Placebo stimulation: duration: 9 seconds, intensity: 2 mA; localisation cerebellum;

SUMMARY:
The purpose of this study is to determine whether transcranial cathodal direct current stimulation (tDCS) delivered over the cerebellum can improve essential tremor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 65 years
* Important essential tremor (bilateral postural and/or action tremor since more than one year)
* Normal physical and neurological examination, except for essential tremor
* Insufficient efficiency of usual essential tremor's treatment
* No treatment altering the cortical excitability
* Agreement to use a medically acceptable method of contraception throughout the study for female of childbearing potential
* mini-mental status score >24

Exclusion Criteria:

* Age < 18 years and > 65 years
* Current neurological or psychiatric illness other than essential tremor
* Individual who is on medication which is known to lower seizure threshold
* Previous history of seizure, loss of conciousness or current active epilepsy
* Contraindication for MRI or TMS study
* Intake of antiepileptic medications for essential tremor (barbiturates, gabapentine, topiramate, clonazepam), within the 7 days preceeding the first visit
* alcohol intake within the 24 hours preceeding the first visit
* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control
* Individual who have MMS ≤ 24/30 or patients legally protected or inability to provide an informed consent
* Simultaneous participation in another clinical trial
* Patients who are not enrolled at social security

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in tremor amplitude on clinical rating scale | 10 minutes after the end of tDCS

SECONDARY OUTCOMES:
Change from baseline in tremor amplitude on accelerometric recording | During tDCS, 10 mn, 60 mn and 90 mn after the end of tDCS
Change from baseline in tremor amplitude on electromyographic recordings | During tDCS, 10 mn, 60 mn and 90 mn after the end of tDCS
Change from baseline in tremor amplitude on digitized tablet | During tDCS, 10 mn, 60 mn and 90 mn after the end of tDCS
Change from baseline in tremor amplitude on clinical rating scale | During tDCS, 60 mn and 90 mn after the end of tDCS
Change from baseline of amplitude of motor evoked potentials elicited by TMS | 10 mn, 60 mn and 90 mn after tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Flamand-Roze, MD, Principal Investigator — Institut du Cerveau et de la Moelle et Fédération de Neurologie de l'Hôpital Pitié-Salpétrière, Paris
Locations (1):
- Institut du Cerveau et de la Moelle, Hôpital Pitié-Salpétrière, Paris, France